CLINICAL TRIAL: NCT05047822
Title: Real-world Effectiveness of the Oxford/AstraZeneca COVID-19 Vaccine in England. An Observational Retrospective Cohort Study Using Secondary Databases to Establish Effectiveness of the Oxford/AstraZeneca COVID-19 Vaccine in England.
Brief Title: Oxford/AstraZeneca COVID-19 Vaccine Effectiveness in England
Acronym: RAVEN
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: The Chancellor, Masters and Scholars of the University of Oxford (Unknown)
Responsible Party: Sponsor
Other Study IDs: D8111R00007
Record Dates: First submitted 2021-08-27; First posted 2021-09-17 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Covid-19 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Concurrent Controls
- Vaccinated Cohort

SUMMARY:
This is a retrospective cohort study to assess the real world effectiveness of the Oxford/AstraZeneca COVID-19 vaccine in England. The study is using linkage of the English national databases on COVID-19 vaccination, testing, medical records, hospitalization, and death.

DETAILED DESCRIPTION:
The United Kingdom (UK) is one of the first countries that introduced a mass vaccination campaign for COVID-19 and vaccination of the adult population first focused on the oldest age groups, their carers and health care workers (JCVI, 2020). Three COVID-19 vaccines were licensed and are being used including the Moderna, the BioNTech/Pfizer, and the Oxford/AstraZeneca vaccines. Vaccination with the BioNTech/Pfizer vaccine started in December 2020 and the Oxford/AstraZeneca vaccine started in early January 2021. This study is to primarily assess the effectiveness of the Oxford/AstraZeneca COVID-19 vaccine. Given the known high efficacy of the mRNA vaccines in randomized controlled trials (RCTs) and real-world evidence studies, the study aims also to evaluate the vaccine effectiveness (VE) of other COVID-19 vaccines as a validation of the study's methods. On 16 September 2021 it was announced that Booster doses would be introduced in the UK to address vaccine waning and for groups with a suboptimal response. Little is known about health care resource utilisation (HCRU) and health care costs for those who have had COVID-19 or by individual clinical risk group. The RAVEN study is a retrospective cohort study to assess the real-world effectiveness of the Oxford/AstraZeneca COVID-19 vaccine in England. The study is using linkage of the English national databases on COVID-19 vaccination, testing, medical records, hospitalization, and death. Analyses will examine the effectiveness of one and two doses, and booster or other additional doses if applicable. This study's extension (October 2021) adds a more detailed exploration of VE in risk groups and an evaluation of the HCRU by people with COVID-19 compared with those who are vaccinated.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for any COVID-19 vaccination based on age at index date
* Have continuous data coverage for the COVID-19 infection datasets
* Have continuous data coverage in other linked databases for a minimum of 12 months prior to the index date

Exclusion Criteria:

• People with a history of COVID-19 infection (confirmed by reverse transcriptase polymerase chain reaction (RT-PCR) or not) prior index date

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 12 years old or older population in England who met inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 18373714 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Incidence rate of COVID-19 related hospitalizations, COVID-19 related ICU admissions and COVID-19 related deaths | up to 12 months

SECONDARY OUTCOMES:
Incidence rate of all-cause hospitalisations, all-cause ICU admissions and all-cause deaths | up to 12 months
Incidence of positive SARS-CoV-2 test | up to 12 months
Incidence of medically attended COVID-19 | up to 12 months
Incidence of COVID-19 related emergency department visit | up to 12 months
COVID-19 related healthcare resource utilisation | up to 12 months
  Number of primary care consultations, prescriptions, medical tests and investigations, hospital outpatient attendances and procedures, hospital emergency department attendances without admission, hospital admissions
Costs for COVID-19 related healthcare | up to 12 months
  Costs for primary care consultations, prescriptions, medical tests and investigations, hospital outpatient attendances and procedures, hospital emergency department attendances without admission, hospital admissions

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Leeds, United Kingdom

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8111R00007&attachmentIdentifier=242daf89-4ffb-4fbe-ba79-f05ed679b563&fileName=CSR_Synopsis_Final_16Oct_all_Redacted.pdf&versionIdentifier=